CLINICAL TRIAL: NCT06875518
Title: Comparative Study of Blood Loss in Total Laparoscopic Hysterectomy by Ligation the Uterine Arteries in Different Techniques.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mostafa Bahaa (Other)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Lecturer, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 8749
Record Dates: First submitted 2025-03-09; First posted 2025-03-13 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Group 1 (BTLH with bilateral uterine artery ligation from its origin): The round ligament close to the pelvic side wall is first coagulated and separated before the procedure is applied.
  Interventions: Procedure: BTLH with bilateral uterine artery ligation from its origin
- Conventional TLH (Active Comparator): The conventional TLH technique involved division of the corneal pedicles and securing the uterine pedicles. Preoperative Preparation of bowel wasn't routinely done to improve enhanced recovery of patients.
  Interventions: Procedure: Conventional TLH

INTERVENTIONS:
Procedure: BTLH with bilateral uterine artery ligation from its origin — The round ligament close to the pelvic side wall is first coagulated and separated before the procedure is applied. Further incision is then made in the peritoneum. The bladder fold is pulled downward by opening the anterior leaf of the wide ligament. It shows the ureters lateralized and the posterior leaf of the wide ligament. After that, the ureters' path is shown, the retroperitoneal area is revealed, and the location where the uterine artery leaves the iliac artery is seen.
  Arms: Control group
Procedure: Conventional TLH — The conventional TLH technique involved division of the corneal pedicles and securing the uterine pedicles. Preoperative Preparation of bowel wasn't routinely done to improve enhanced recovery of patients. Antibiotic prophylaxis with 3rd generation cephalosporin and metronidazole was given one hour preoperatively. Obese patients received subcutaneous low molecular weight heparin and compression devices after surgery. Under general anesthesia, patients were placed in a Lloyd Davis position.
  Arms: Conventional TLH

SUMMARY:
Following Caesarean section, hysterectomy is the second most common major gynecological surgery, with approximately 600,000 procedures performed annually in the USA. Since Reich et al. first reported a total laparoscopic hysterectomy (TLH) in 1989, numerous studies have confirmed its feasibility and reproducibility. Evidence increasingly supports TLH over vaginal hysterectomy (VH) and total abdominal hysterectomy (TAH) for benign gynecological conditions. The development and rapid advancement of laparoscopic instruments and techniques have enabled the safe and successful completion of complex procedures using minimally invasive approaches. Women with a higher BMI or requiring complex surgeries benefit from reduced postoperative complications with laparoscopic operations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 35-60 years Patients presented with menometrorrhagia unresponsive to medical treatment, and uterine pathology such as adenomyosis or multiple fibroids.

Exclusion Criteria:

* Patients were excluded if they had: medical conditions preventing pneumo-peritoneum
* Patients with medical conditions hindering proper ventilation during general anesthesia.
* Patients diagnosed with endometrial carcinoma and patients with uterine size larger than 24 weeks were excluded.
* Patients with excessive adhesions precluding access to the uterine arteries were not enrolled in the study.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Intra operative blood loss | 24 hours
  Vaginal vault is identified and cut laparoscopically using monopolar hook over the manipulator cup and bipolar grasper for hemostasis until the specimen is detached completely. The uterus with cervix is delivered vaginally. The vaginal vault is sutured laparoscopically with number 1 delayed absorbable suture (Polyglactin; vicryl).
  The total blood loss is calculated from the suction apparatus.

CONTACTS AND LOCATIONS:
Locations (1):
- Mostafa Bahaa, Damietta, New Damietta, Egypt